CLINICAL TRIAL: NCT04885582
Title: The Relationship Between HLA Tissue Compatibility and Biliary Complications in Patients With Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ersin Gündoğan, Assoc Prof, Inonu University
Other Study IDs: 2017/133
Record Dates: First submitted 2021-05-11; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Liver Transplant; Complications; HLA Antigens
Keywords: Liver Transplant; Complications; HLA; biliary fistula; biliary stricture
MeSH Terms: conditions — Biliary Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with biliary complications: patients with postoperative biliary fistula, biliary stenosis
  Interventions: Other: HLA antigen results
- Patients without biliary complications: patients without postoperative biliary fistula and biliary stenosis
  Interventions: Other: HLA antigen results

INTERVENTIONS:
Other: HLA antigen results — HLA-A, HLA-B, HLA-DR tissue matching results in both groups will be compared.

SUMMARY:
Liver transplantation has become the accepted treatment option for advanced liver failure in recent years. In addition to the increase in the number of centers performing transplant and the decrease in complication rates depending on the experience gained, the most common biliary complications did not improve at the desired level. For this reason, studies in this field are frequent today.

The structural complexities of HLA antigens have been the subject of investigation in recent years. With the development of DNA and RNA amplification methods; It is increasingly difficult for physicians to keep up with the increasing burden of knowledge regarding the genetic aspects of these antigens. Concrete benefits of this gene complex, which has been investigated in various fields and preserves its mystery, have not been determined in liver transplant patients. However, there are publications showing its connection with the bile epithelium in liver transplantation and its relationship with the disappearing bile duct syndrome. In this study, our aim is to explain whether the bile duct complications, which appear like a continuous wall and can lead to frightening pictures, are related to HLA tissue compatibility.

ELIGIBILITY:
Inclusion Criteria:

* patients with liver transplantation and tested for HLA antigen (recipient - donor)

Exclusion Criteria:

* patients who died early Patients whose HLA antigen is not checked

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had liver transplantation and HLA tissue tests between 2017 and 2019 at Inonu University liver transplant institute
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Bliary complications | 2 years
  Biliary fistüla, biliary stenosis

CONTACTS AND LOCATIONS:
Locations (1):
- Health science University - Kayseri State Hospital, Kocasinan, Kayseri, Turkey (Türkiye)